CLINICAL TRIAL: NCT07308171
Title: Nasal Airflow to Modulate Dyspnea in Tracheostomized Patients
Acronym: MODUS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP251423
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Ventilated Patients
Keywords: Mechanical ventilation; Tracheostomy; Nasal stimulation
MeSH Terms: interventions — BaseLine dental cement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients ventilated (Experimental): Baseline ventilator settings under pressure support
  Interventions: Procedure: Baseline; Procedure: Installation of high flow humidified air cannula; Procedure: Nasal air puffs; Procedure: propeller fan (FAN)

INTERVENTIONS:
Procedure: Baseline — patient ventilated through the tracheostomy with initial ventilator settings
Procedure: Installation of high flow humidified air cannula — Installation of high flow humidified air cannula with inspired oxygen fraction (FiO2) 21%
Procedure: Nasal air puffs — Nasal air puffs synchronized with the inspiratory time of the ventilator
Procedure: propeller fan (FAN) — Stand-alone fan at the bedside directed toward the face of the patient

SUMMARY:
The hypothesis of the present study is that restoring nasal stimulation alleviates dyspnea and improves respiratory drive. The aim of this study is to compare three non-pharmacological approaches designed to restore nasal stimulation (continuous nasal airflow, nasal sprays, and facial airflow) in tracheotomized patients dependent on mechanical ventilation.

DETAILED DESCRIPTION:
Nasal stimulation is generated by breathing, which enables olfaction and helps to rhythm brain activity. The loss of nasal stimulation in tracheotomized patients who are dependent on mechanical ventilation may negatively affect respiratory drive and contribute to dyspnea. Restoring nasal airflow therefore emerges as an attractive non-pharmacological approach to treat dyspnea in patients undergoing mechanical ventilation weaning.

The hypothesis of the present study is that restoring nasal stimulation alleviates dyspnea and improves respiratory drive. The aim of this study is to compare three non-pharmacological approaches designed to restore nasal stimulation (continuous nasal airflow, nasal sprays, and facial airflow) in tracheotomized patients dependent on mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Tracheostomy and mechanical ventilation
3. Dyspnea ≥3
4. Consent to participate
5. Affiliation to health insurance

Exclusion Criteria:

1. Agitation, delirium
2. Continuous use of sedatives
3. Patients under law protection
4. Inmates
5. Patients without health insurance
6. Breastfeeding and pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Dyspnea | minute 20
  visual analogical scale

SECONDARY OUTCOMES:
airway occlusion pressure | minute 20
  visual analogical scale
end expiratory occlusion pressure | minute 20
  visual analogical scale
respiratory electromyogram (EMG) | minute 20
  visual analogical scale
tolerance | minute 20
  visual analogical scale

CONTACTS AND LOCATIONS:
Overall Officials: Martin Dres, MD PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.